CLINICAL TRIAL: NCT02131168
Title: Investigating the Epidemiology of Inflammatory Bowel Disease in Hong Kong: An Inception Cohort and Follow up Study (IBD EPI Study)
Brief Title: Epidemiology of IBD in Hong Kong: An Inception Cohort and Follow up Study
Acronym: ACCESS
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: IBD EPI
Record Dates: First submitted 2014-04-29; First posted 2014-05-06 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — One stool sample will be collected for microbiology tests 10 ml of blood will be stored for genetic analysis
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Crohn's disease and ulcerative colitis are inflammatory disorders of the gut which cause major life-long disability. They affect males and females, with the commonest age of onset in childhood, teens and early adult life. Previously restricted almost exclusively to the West, these conditions are becoming much more common in Asian countries, including Hong Kong - the cause of this dramatic change is unknown.

The cause of IBD is widely accepted as relating to the mucosal immune response to stimulation from the gut bacteria, on a background of genetic susceptibility. The bacteria and other organisms in the gut play a central role in the development of IBD in the West. However it is unknown if the gut bacteria differ between Chinese patients with IBD and non-IBD (healthy subjects) in Hong Kong, and whether it is affected by diet or changes in diet. A family history is the largest risk factor for the disease. More than 50 different genes associated with IBD have recently been identified in the West and preliminary data showed that Chinese patients have a different genetic profile to Western populations.

This project aims to explore the true incidence of IBD in Hong Kong and factors that may be contributing to, or causing, the increase of IBD in Hong Kong. Investigators aim to investigate the number of new cases of IBD within a five year period and factors that may account for the cases. Investigators will also study the choice of medical therapy, quality of life and quality of health care in patients with IBD.

DETAILED DESCRIPTION:
Investigators will create the first web-based Hong Kong inception cohort database. Via the web registration investigators intend to form a new prospective, uniformly diagnosed, population-based inception cohort of patients with IBD. Physicians, gastroenterologists, family doctors, surgeons and pathologists in our study area will be notified repeatedly about the study by letter, telephone, internet, personal visit of the investigators, and encouraged to inform investigators of every possible new case of IBD (persistent or relapsing diarrhoea, blood and/or mucus in the stools for more than three weeks, or abdominal pain and weight loss). Endoscopic, pathology and radiology records will be canvassed repeatedly for likely cases, both electronically and manually. By these methods investigators intend to capture over 90% of possible cases. New patients will be included during a five-year period, 01.04.2011 - 31.03.2016, followed by a five year follow-up period until 31.03.2021. All patients are required to meet the diagnostic criteria for IBD on the basis of clinical symptoms, endoscopic or radiological evidence or mucosal biopsies. Infectious gastroenteritis, tuberculosis, entamoeba and cancer have to be ruled out. The web-based Database application will be used for online registration of the various registration forms and questionnaires (see list of additional materials), and the database is located on a central secured server.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed IBD patients based on clinical, endoscopic, histologic or radiologic criteria will be included during the study period

Exclusion Criteria:

* Any patients with a diagnosis of tuberculosis, infectious enteritis, amebiasis, or GI cancer that may mimic the diagnosis of IBD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed IBD patients in the local area
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Number of new cases of IBD | Up to 5 years
  Data of new IBD case will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No